CLINICAL TRIAL: NCT05954156
Title: Clinical Performance of Injectable Resin Composite Versus Dual Cured Resin Cement For Cementation of Indirect Hybrid Ceramic Onlay Restorations: A Randomized Clinical Trial
Brief Title: Injectable Resin Composite Versus Dual-cured Resin Cement for Cementation of Indirect Onlay Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hamsa Ashraf Abd El Menam, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRS_DCRC
Record Dates: First submitted 2023-07-05; First posted 2023-07-20 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cementation Teeth; Badly Broken Down Vital Teeth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injectable restorative resin composite material used for cementation (Experimental): Highly filled injectable composites display properties in a manner similar to resin cements due to their unique viscosities. This with the added benefits of higher filler content, thus improved mechanical and physical properties with the easy placement and handling properties which can improve clinical performance and durability of indirect restorations. (Fugimoto et al., 2019)
  Interventions: Other: Injectable restorative resin composite
- Dual cured resin cement (Active Comparator): Dual cured resin cement is chosen as a comparator (gold standard )for the cementation of indirect restorations. (Sadighpour et al., 2018) Resin cement is insoluble and has superior mechanical and physical properties, compared with other previous luting materials. The clinical advantages of resin cement include high resistance to compression forces, low thermal expansion coefficients, high flexural strengths, and hardness. In addition, resin cement is characterized by adhesion to many materials, the ability to modify shade and color, high retention, resistance to wear at the margin of the restoration, and low marginal permeability. Resin cement provides optimal bond with resin composite indirect restorations and evenly distributes the compression force along all contact surfaces. (Gurdal et al., 2018
  Interventions: Other: Dual cured resin cement

INTERVENTIONS:
Other: Injectable restorative resin composite — The introduction of injectable composites, according to available literature, offers a simple and efficient solution for the cementation of veneers. This versatile, injectable restorative composite unites easy handling, high physical properties and excellent aesthetics. Generally used as a restorative material, it can also be used for the cementation of veneers and some inlays/onlays, thus considered as good alternative to preheated composite. (Alajrash MM et al., 2020)
  Arms: Injectable restorative resin composite material used for cementation
Other: Dual cured resin cement — Resin cements are widely used due to their strong adhesion, and compatibility with various restorative materials, including ceramics and zirconia. They bond to enamel and dentin through functional monomers such as MDP, and 4-META, forming a stable hybrid layer. Based on their bonding mechanism, resin cements are classified as adhesive or self-adhesive, while their polymerization method -chemical, light, or dual-cure-allows for versatility in clinical applications
  Arms: Dual cured resin cement

SUMMARY:
Marginal integrity is considered the main essential part of indirect restorations and any discrepancy after cementation and poor marginal fit can lead to microleakage, marginal discoloration, dissolution of cement and secondary caries. The type of cement used plays an important role and can govern the amount of augmentation in discrepancy after cementation.

Although resin cement is still the gold standard luting agent for the cementation of all indirect restoration, it lacks some properties that may be available in the restorative resin composite such as higher filler loading, higher mechanical properties and wear resistance.

may have been the first to propose the use of restorative, flowable resin composite as a luting agent for ceramic inlays. These authors demonstrated that with respect to polymerization rate, there were no advantages of dual curing-resin compared to light curing only. In addition, the overall handling of the light-curing flowable restorative resin composite was judged to be easier than that of the dual cured material. The same conclusions were drawn by Kramer and franken Berger who added that less luting resin composite overhangs were found with the light polymerized composite-resin because the clinician has more time for excess removal prior to polymerization. The claimed further potential advantages of using restorative rein composite as a luting agent is their resistance to wear which proved to be superior to resin cements

DETAILED DESCRIPTION:
the author presented a review on the updates of dental cements, focusing on the composition, properties, advantages, limitations, and indications of the various cements available. Nowadays, dental restorations are made from various biomaterials, and depending on each clinical case, an appropriate luting material will be selected. There is no luting material that can be universally used. Therefore, it is important to distinguish the physical, mechanical, and biological properties of luting materials in order to identify the best options for each case. Nowadays, the most commonly used dental cements are glass-ionomer and resin cement. The type, shade, thickness of resin cement and the shade of the ceramic, all together, have a tangible influence on the final restoration color. Surface treatments of the restoration increase the micro tensile bond strength. Hence, the proper surface treatment protocol of both the substrate and restoration surfaces is needed before cementation. Additionally, the manufacturer's instructions for the thin cement-layer thickness are important for the long-term success of the restoration.

the author conducted a study to evaluate the performance of two different adhesive resin cement systems in the cementation of inlay/onlay restorations produced from resin nanoceramic blocks using the CAD/CAM system. The methodology was total of 70 inlay/onlay restorations made from Cerasmart (GC, Tokyo, Japan) resin nanoceramic blocks using CEREC Omnicam (Sirona Dental, Bensheim, Germany) were placed in 53 patients. The restorations were cemented with RelyX U200 Automix (3M ESPE, Seefeld, Germany) self-adhesive resin cement (RXU) after selective enamel etching or with G-CEM LinkForce (GC, Tokyo, Japan) adhesive resin cement (GCL) in combination with a universal adhesive (G-Premio Bond) in selective etch mode. At baseline and after 6, 12, and 18 months, restorations were examined by two calibrated clinicians according to modified USPHS criteria. . he concluded that the two resin cement systems showed acceptable clinical performance for the cementation of resin nanoceramic CEREC Omnicam inlay

the author conducted a study to evaluate the retention strength of zirconia crowns luted with two types of resin cement under environmental pressure changes.Thirty zirconia crowns were fabricated by using computer-aided design/computer-aided manufacturing (CAD/CAM) system and were cemented by Panavia F2.0 (PAN), hand-mixed RelyX Unicem (UNH), or auto-mix RelyX Unicem Aplicap (UNA) cements on the corresponding extracted human molars. The samples were randomly divided into three groups according to the cement type. After 3000 thermal cycles, the cemented crowns were subjected to 24 pressure cycles (0 to 5 atmospheres). The retention force (N) of the specimens was measured in a universal testing machine. To normalize the retentive force, the recorded force was divided by the surface area of each tooth for measuring the retentive strength (MPa). he concluded that. The adhesive failure mode was predominant in all the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vital, asymptomatic, badly broken-down lower molar exhibiting at least two missing walls and one or more weakened or absent cusps (indicated for an onlay restoration), classified as ICDAS score (5)
* Patients with at least 20 teeth under occlusion.
* Age: 20-40 years.
* Males or females.
* Co-operative patients approving to participate in the trial.
* Good oral hygiene measures
* Teeth with no signs of pulpal involvement; healthy periodontal status; favorable occlusion
* Those in good general health.

Exclusion Criteria:

* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis or periapical pathosis
* Teeth supporting removable prostheses, or orthodontic appliances.
* Candidates with parafunction or bruxism or temporomandibular joint disorders
* Candidates with systemic diseases or disabilities that may affect participation.
* Heavy smoking.
* Pregnancy.
* Lack of compliance.
* Severe or active periodontal disease
* Non-vital or endodontically treated teeth
* Xerostomia
* Drug addiction; or any condition that could compromise study compliance.

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Clinical Performance | 18 months change from baseline to 6, 12, and 18 months
  Retention, marginal integrity, secondary caries, anatomic form, surface texture, proximal contact and postoperative hypersensitivity. All these outcomes are measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable ,charlie is not accepted

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Ashraf H, El Tannir A, El Zohairy A, Kamal D. Clinical performance of indirect hybrid ceramic onlay restorations cemented with injectable resin composite versus dual-cure resin cement: an 18-month randomized clinical trial. BMC Oral Health. 2025 Sep 23;25(1):1419. doi: 10.1186/s12903-025-06903-5. PMID 40988059